CLINICAL TRIAL: NCT03854201
Title: Personalized Exercise Counseling to Promote Workability and Health of Municipal Workers With Musculoskeletal Pain in Nokia City, Finland
Brief Title: Personalized Exercise Counseling to Promote Workability
Acronym: PEC-Nokia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: UKK Institute (Other)
Collaborators: City of Nokia (Unknown)
Responsible Party: Principal Investigator, Jaana Suni, Reserach and Development Manager, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKK Institute_Nokia City; ETL code R18184 (Other: Regional Ethics Committee of Tampere University Hospital)
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Physical Functioning; Musculoskeletal Pain; Quality of Life; Physical Activity
Keywords: workability, sickness absence, health promotion, costs
MeSH Terms: conditions — Musculoskeletal Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with two-arm study design:
  1. Intervention-arm: Face-to-face Personalized Exercise Counseling combined with interactive ExSed® accelerometer (PEC)
  2. Non-treament-arm: Participation in the study measurement only, and written information with individual feedback on blood sugar and lipid profile, fitness test results and objectively measured physical activity 24/7 after each of the four measurement points (Control-arm)
Who Masked: Investigator
Masking Description: After the screening phase, all electronic questionnaire data will be collected in the form of pseudonymity i.e. using only the numeric identification codes. All data (results of blood samples, fitness tests, research accelerometers) will be saved and analysed using only the codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Exercise Counseling (PEC) (Experimental): The Personalized Exercise Counselling intervention includes 3 face-face counseling sessions and 4-6 phone calls during six months. In addition, the participants are provided with the ExSed® interactive accelerometer to record their physical activity 24/7 from which they will receive personal daily feedback on their smart phone, which is provided to each person not having a suitable one of their own to be used during the 6-month intervention period.
  Interventions: Behavioral: Personalized Exercise Counseling (PEC)
- Control-arm (No Intervention): The participants only take part in the study measurements at baseline and the three follow-up time points. They will be provided personal written information by the UKK Institute on their blood sugar and lipid profiles, objectively measured physical activity (light, moderate, vigorous), standing, sedentary behaviour and sleep, and the three fitness tests measuring flexibility, muscular strength and cardiorespiratory fitness.

INTERVENTIONS:
Behavioral: Personalized Exercise Counseling (PEC) — At the first counseling appointment, PEC-participants answer the physical activity (PA) questionnaire, perform fitness tests and discuss with their exercise instructor. The target is a personalized short-term PA plan including where and when the PA/exercise takes place and what is the mode. Participants may choose instructed group-exercise sessions provided by the municipal sports/leisure sector or exercising alone as preferred. The exercise instructors utilize the fitness test results and feedback data of the research accelerometers by the UKK Institute to guide the participants. The PEC includes 2 more face-to-face sessions and 4-6 phone calls by the instructors aimed at checking the realization of exercise plans and discussing the outcomes provided by the interactive accelerometer.
  Arms: Personalized Exercise Counseling (PEC)

SUMMARY:
The study design is a 2-arm randomized controlled trial with 6-month intervention period and follow-up at 6, 12 and 24 months among blue-color workers of Nokia City with reduced work ability and high number of musculoskeletal problems. The participants (n=190) will be randomly assigned to intervention-arm providing face-to-face Personalized Exercise Counseling combined with interactive accelerometer (PEC-arm) or a non-intervention Control-arm. The study aims at improving workability (main outcome) and reducing musculoskeletal pain by counseling and motivating the workers to increase physical activity and exercise according to self-selected modes. Exercise instructors of Nokia City are responsible for providing the face-to-face part of PEC. The Urho Kaleva Kekkonen (UKK) Institute is responsible for providing online feedback of the data collected by the interactive ExSed® accelerometer, stored and analyzed in the Cloud, from where the participants in the PEC-arm receive daily feedback thru a smart phone application. Cost-effectiveness of the PEC-intervention compared to the Control-arm in terms of quality adjusted life-years (QALY) and days of sickness absence are also investigated. The following measurements will be taken at baseline and the three follow-up timepoints: work-, health- and physical activity related factors collected by two electronic questionnaires, objective measurements of movement continuum (sleep, sedentary behavior, standing-ups, standing, light activity, moderate activity, vigorous activity) for 24/7 (RM42 research accelerometer), 3 tests of physical fitness and blood samples related to blood sugar and lipid profile.

DETAILED DESCRIPTION:
Sick-leaves due to musculoskeletal disorders (MSDs) among municipal workers of Nokia City increased notably during the year 2017, which was noticed as increased call and burden in occupation healthcare settings. According to the disease grading statistics of early retirement, MSDs were the leading cause. Due to the afore facts Nokia City composed a novel model of co-operation between the personnel administration and exercise facilities of Nokia City: The coordinator of wellbeing (occupational nurse) now prescribes exercise referrals for patients to directly contact the sports sector for personalized exercise counseling.

The purpose of the present study is to investigate the effectiveness and cost-effectiveness of the afore described novel operations model of exercise referral in the Nokia City. Personalized Exercise Counseling (PEC) intervention guides and motivates the workers to set and achieve personal exercise/physical activity goals. The hypothesis is that the PEC improves workability (main outcome) and reduces musculoskeletal pain, and thus improves quality of life and reduces days of sickness absence. Regarding cost-effectiveness of the PEC-arm is expected to be cost-effective in terms of quality adjusted life-years (QALY) and days of sickness absence compared to the Control-arm.

The target population of the PEC-Nokia study is practical nurses, personnel of kitchen and cleaning service and janitorial service. In case that the number of participants fulfilling the inclusion criteria of these occupational groups is not adequate to reach the number needed to be randomized (n=190), other occupations may be recruited.

Sample size was calculated based on the work ability score (WAS) i.e. current work ability compared to lifetime best on numeric rating scale from 0 (completely unable to work) to 10 (work ability at its best). Thus, to detect a difference in main effects (i.e., Personalized Exercise Counselling (PEC) group vs. non-treatment group (Control) with a significance level of 0.05 and a power of 90%, the study required at least 150 participants (75 in each study-arm). For compensation of probable loss of participants to follow-up, the aim is to recruit 190 participants. We expect that there would be a minimal difference of 15% between the PEC-arm and Control-arm among those with improved WAS-score to the good level (i.e. at least 8). We expect that 5% of the participants in the Control-arm and 20% in the PEC-arm will reach the afore target. Reductions of 30% or 15mm (0-100) in intensity of musculoskeletal pain levels at neck-shoulder, lower back, and knee would meet the criteria of clinically important change.

The participants (n=190) will be randomly assigned into 6-month Personalized Exercise Counseling combined with interactive accelerometer (PEC-arm) or a non-intervention Control-arm. Statistician KT will randomly assign about 200 persons to one of the two parallel groups in a 1:1 ratio using a computer-generated procedure. The codes of the study group will be provided to the participants fulfilling the inclusion criteria, using the method of sealed envelopes, immediately after the person has given his/her written consent to participate to the well-being coordinator (specialist nurse of occupational health employed by Nokia City). Only the investigators (i.e. the research group) will be blinded to group allocation.

Electronic questionnaires have been prepared to cover the following: Work-related factors include perceived physical strain, perceived exertion after typical work day at different body sites of musculoskeletal structures and work stress; Health-related factors include perceived health, depression, sleep and recovery, quality of life and days of sickness absence; Physical activity related factors include preferred activity modes and motivation, Fear Avoidance Beliefs related to physical activity at work and leisure-time. In addition, the following physical tests will be used to measure health-related fitness: Neck-shoulder mobility for flexibility, Modified push-ups for upper body strength and trunk stability and 6 minutes' walk test for cardiorespiratory fitness in terms of distance walked and predicted maximal oxygen uptake.

ELIGIBILITY:
Inclusion Criteria:

• Reduced workability of less than 8 in the numeric rating scale assessed by the Work Ability Scale (WAS), an item of the Work Ability Index (WAI), as "Current work ability compared with lifetime best rated on a numeric rating scale from 0 (completely unable to work) to 10 (work ability at its best)"

Exclusion Criteria:

• not likely to be albe to do one's current job two years from now assessed with Future Walk Ability (FWA) item from WAI "Do you believe that, from your health perspective, you will be able to do your current job two years from now?"' was rated with three response alternatives: unlikely (1), not certain (2) and relatively certain (3)

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in Work ability score (WAS) at follow-up time points | Baseline, 6, 12 and 24 months
  Current work ability compared with lifetime best rated on a scale from 0 (completely unable to work) to 10 (work ability at its best).

SECONDARY OUTCOMES:
Intensity of musculoskeletal pain measured with Visual Analog Scale (VAS) in different anatomical sites: neck-shoulder, lower back, upper extremities, lower extremities | Baseline, 6, 12 and 24 months
  100-mm visual analog scale, 40mm indicating clinically meaningful level of pain
Objectively measured physical activity continuum (24/7) for 7 days | Baseline, 6, 12 and 24 months
  During waking hours the small size three axial research accelerometer RM42 is worn on the right waist in an elastic belt; during sleeping hours in a wrist
Cost effectiveness: Quality Adjusted Life Years (QALY) | Baseline, 6, 12 and 24 months
  Cost-effectiveness is expressed as incremental cost-effectiveness ratios (ICERs), calculated as the ratio of the difference in mean total costs (including healthcare costs, medication, costs of sickness absence, and intervention costs) and main effects (i.e., change in QALY) at the level of the study-arms.
  QALY were calculated from the SF-6D score derived from the original SF-36 data, which is a validated instrument for measuring the physical and mental components of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Erkkilä, Dr., Study Chair — Human Reserach Manager, City of Nokia
Locations (1):
- UKK Insitute for Health Promotion Research, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No